CLINICAL TRIAL: NCT03739099
Title: Assessment of the Efficacy of Closed-loop Insulin Therapy (Artificial Pancreas) on the Control of Type 1 Diabetes in Prepubertal Child in Free-life: Comparison Between Nocturnal and 24-hour Use on 18 Weeks, Followed by an Extension on 18 Weeks
Brief Title: Efficacy of Closed-loop Insulin Therapy in Prepubertal Child in Free-life
Acronym: FREELIFE-KID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF 7580
Record Dates: First submitted 2018-11-05; First posted 2018-11-13 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes Mellitus in Prepubertal Children
Keywords: Type 1 diabetes; Prepubertal children; Closed-loop insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed-loop insulin delivery 24/7, day and night (Active Comparator): Closed-loop subcutaneous insulin infusion driven by continuous glucose monitoring through an algorithm
  Interventions: Device: Closed-loop insulin infusion driven by continuous glucose monitoring through an algorithm, in free-life conditions
- Closed-loop insulin delivery 7/7, dinner and night (Other): Closed-loop subcutaneous insulin infusion driven by continuous glucose monitoring through an algorithm
  Interventions: Device: Closed-loop insulin infusion driven by continuous glucose monitoring through an algorithm, in free-life conditions

INTERVENTIONS:
Device: Closed-loop insulin infusion driven by continuous glucose monitoring through an algorithm, in free-life conditions — Continuous subcutaneous insulin infusion according to an automated algorithm from continuous glucose monitoring data
  Other Names: Artificial pancreas

SUMMARY:
The study is a randomized trial preceded by a run-in period and followed by a non-randomized study extension. After 3 weeks of outpatient use of study pump (1 week) and study pump+CGM (2weeks) as run-in period, patient and parents will be admitted for 4-hour training to closed-loop (AP) mode. Following randomization (1:1), patient will be allocated to '24-hour' use of AP or 'dinner and overnight AP mode/day time pump and CGM use' for the next 18-week period. At 18-week visit, a study extension for a further 18-week period will be initiated. AP mode that will be prescribed to all patients will depend from an independent DSMB decision based upon study safety data collected after 6 and 12 weeks from the first 30 included patients. Visits will occur at week 27 (safety follow-up) and 36 (final visit).

DETAILED DESCRIPTION:
The study is a randomized trial preceded by a run-in period and followed by a non-randomized study extension. After 3 weeks of outpatient use of study pump (1 week) and study pump+CGM (2weeks) as run-in period, patient and parents will be admitted for 4-hour training to closed-loop (AP) mode. Following randomization (1:1), patient will be allocated to '24-hour' use of AP or 'dinner and overnight AP mode/day time pump and CGM use' for the next 18-week period. A hotline phone number will be given to the patient and parents so that they can contact the study staff as needed. A logbook will be provided to collect details about hypoglycemic and hyperglycemic episodes, physical activity and noticeable events. Phone calls will be scheduled between investigator and patient+parents 48 hours, 1 week and 2 weeks after AP mode initiation. Potential misbehaviors will be corrected and all questions answered. If needed, AP parameters may be revised and reconfigured. Hospital visits will be scheduled 6, 12 and 18 weeks after AP mode initiation for the same purposes, plus HbA1c measurement at week 12 and 18. At 18-week visit, a study extension for a further 18-week period will be initiated. AP mode that will be prescribed to all patients will depend from an independent DSMB decision based upon study safety data collected after 6 and 12 weeks from the first 30 included patients. Visits will occur at week 27 (safety follow-up) and 36 (final visit).

ELIGIBILITY:
Inclusion Criteria:

* Treatment of diabetes by insulin pump since > 6 months
* HbA1c level < 10%

Exclusion Criteria:

* Unwillingness of one parent or the legally responsible party to participate in insulin treatment
* Any associated chronic disease or therapy (except insulin) affecting glucose metabolism

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2022-09-05 (Estimated); Study Completion 2023-05-05 (Estimated)

PRIMARY OUTCOMES:
Percent of time spent in the 70-180 mg/dl glucose range assessed on daily CGM data | 18 weeks
  % time blood glucose in 70-180 mg/dl range

SECONDARY OUTCOMES:
Percent of time spent with glucose level < 70, 60 and 50 mg/dl, assessed on daily CGM data | 18 and 36 weeks
  Percent time while blood glucose is kept in safe 70-180 mg/dl range
Percent of time spent with glucose level > 180 and 300 mg/dl, assessed on daily CGM data | 18 and 36 weeks
  Percent time while blood glucose is kept in safe 70-180 mg/dl range
Percent of time spent in the 70-140 mg/dl glucose range assessed on daily CGM data | 18 and 36 weeks
  Percent time while blood glucose is kept in safe 70-180 mg/dl range
Mean glucose level assessed on daily CGM data | 18 and 36 weeks
  CGM data will be used to calculate daily glucose mean to assess the efficacy of the algorithm on glucose control.
HbA1c level measured at week 12, 18, 27 and 36 | 12,18, 27 and 36 weeks
  Levels of glycated hemoglobin will be measured at different time intervals to assess the clinical impact of the use of the algorithm on patient diabetes.
Number of needed interventions by the patients or care providers to treat hypoglycemia | 18 and 36 weeks
  A logbook will be used all along the study by patients to record carbs intake in case of hypoglycemia. If patient required further assistance, care provider who will record third parties intervention.
Percent of time with AP functional, discriminating between each component failure modes | 18 and 36 weeks
  Percent time while blood glucose is kept in safe 70-180 mg/dl range
Score of the Artificial Pancreas Acceptance Questionnaire | 18 and 36 weeks
  This questionnaire consists of 15 affirmations about the use of AP and patient can answer in a scale from 0 (do not agree) to 6 (totally agree). The global score is calculated by the sum of all answers. A high score means a good acceptation of the system. There is no subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M RENARD, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coutant R, Bismuth E, Bonnemaison E, Dalla-Vale F, Morinais P, Perrard M, Trely J, Faure N, Bouhours-Nouet N, Levaillant L, Farret A, Storey C, Donzeau A, Poidvin A, Amsellem-Jager J, Place J, Quemener E, Hamel JF, Breton MD, Tubiana-Rufi N, Renard E. Hybrid Closed Loop Overcomes the Impact of Missed or Suboptimal Meal Boluses on Glucose Control in Children with Type 1 Diabetes Compared to Sensor-Augmented Pump Therapy. Diabetes Technol Ther. 2023 Jun;25(6):395-403. doi: 10.1089/dia.2022.0518. Epub 2023 Apr 6. PMID 36927054